CLINICAL TRIAL: NCT07009756
Title: Impact of Dietary Supplementation With Cricket Powder on Intestinal Microbiota and Cholesterol Metabolism
Brief Title: How Cricket Powder Affects Gut Microbiome and Cholesterol Metabolism
Acronym: CricketOnME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MU-MOU 2023-334.2710; MU-MOU 2023-334.2710 (Other: Mahidol University)
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hypercholesterolemia
Keywords: gut microbiome; hypercholesterolemia; cricket; insect
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricket Powder First, Then Placebo (Experimental): Participants in this arm will consume a daily serving of cricket powder congee for 21 consecutive days, followed by a 28-day washout period, and then consume a daily serving of placebo congee (pork congee) for another 21 consecutive days.
  Interventions: Dietary Supplement: Cricket Powder; Other: Placebo
- Placebo First, Then Cricket Powder (Experimental): Participants in this arm will consume a daily serving of placebo congee (pork congee) for 21 consecutive days, followed by a 28-day washout period, and then consume a daily serving of cricket powder congee for another 21 consecutive days.
  Interventions: Dietary Supplement: Cricket Powder; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cricket Powder — The intervention product is each serving of cricket powder, which contains 21.5 grams of house cricket (Acheta domesticus) powder blended with pumpkin powder, packed in a sachet. The powder is prepared under sterile conditions and heat-treated to ensure microbiological safety, in compliance with Thai public health regulations.
  Each serving of cricket powder will be consumed together with 32 grams of instant pork-flavored congee, serving as the food base.
  This intervention is distinguished by its use of whole cricket powder as a natural, food-based source of protein, chitin, and bioactive compounds, rather than isolated nutrients or supplements. Unlike many clinical studies that use encapsulated insect protein, purified chitin, or insect extracts, this study utilizes a whole-food approach, incorporating cricket powder into a culturally relevant format, congee, to reflect real-life dietary practices.
Other: Placebo — 32 grams of instant pork-flavored congee that does not contain cricket powder

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death worldwide, including in Thailand. One of the major risk factors for CVD is dyslipidemia, or abnormal levels of cholesterol and other fats in the blood. Recent research suggests that the balance of gut microbiota, the community of microorganisms living in the digestive system, may play a key role in regulating cholesterol levels and overall metabolism.

This study explored the potential health benefits of cricket powder, a high-protein food that is already safely consumed in many parts of the world. Previous studies have shown that cricket powder may increase the number of beneficial gut bacteria, especially Bifidobacterium animalis, which supports the production of short-chain fatty acids (SCFAs) known to improve fat metabolism.

Although crickets are considered safe to eat, more research is needed to understand their effects on gut health and blood cholesterol, especially in people with high cholesterol levels. This study assessed the safety of cricket powder consumption and whether it can help improve gut microbiota balance and lower cholesterol in Thai adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, aged in the 20 - 60 range
* BMI (Body Mass Index) in the range of 18.5 - 29.9 kg/m2
* No underlying diseases
* No gastrointestinal surgery
* The fasting blood parameters of total cholesterol and LDL-C are higher than 200 mg/dL and 130 - 189 mg/dL, respectively.
* The fasting blood triglyceride must be less than 500 mg/dL.
* The fasting blood glucose must be less than 110 mg/dL.
* ALT (Alanine aminotransferase) and AST (Aspartate aminotransferase) must be less than 60 units/L.
* eGFR (estimated glomerular filtration rate) must be at least 90 mL/min/1.73 m2.
* Blood pressure must be less than 160/90 mmHg.
* Heart rate must be less than 100 times/minute.
* No smoking
* Be able to consume pork congee

Exclusion Criteria:

* Allergic to insects, chitin, chitosan, shrimp, dust mites, and other crustacean products
* Pregnant or breastfeeding
* Participating in other research projects, and receiving drugs, herbs, and supplements
* Receiving steroid, antibiotic, or other drugs that may affect lipid metabolism
* Consuming alcohol more than 2 drinks per day e.g., beer of 24 ounces, wine of 10 ounces, and distilled spirits of 3 ounces
* Regularly consuming probiotic products and cannot stop consuming them
* Having histories of diabetes, chronic liver diseases, chronic kidney diseases, cardiovascular diseases, cancer, anemia, irritable bowel syndrome, ulcerative colitis, or anaphylaxis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Gut Microbiota Composition | 70 days
  Assessed by analyzing stool samples using 16S rRNA gene sequencing to evaluate changes in the relative abundance and diversity of gut microbiota
Short-Chain Fatty Acid (SCFA) Profiles | 70 days
  Quantification of fecal SCFA concentrations (e.g., acetate, propionate, and butyrate) using gas chromatography and metabolomic analysis to assess microbial metabolic activity and functional output

SECONDARY OUTCOMES:
Change in Blood Lipid Levels | 70 days
  Measurement of serum lipid profiles, including total cholesterol, LDL-C, HDL-C, and triglycerides, to evaluate the effect of cricket powder on lipid metabolism
Adverse Events and Safety Monitoring | 70 days
  Assessment of adverse effects through participant self-report, clinical observation, and relevant laboratory parameters to evaluate the safety of daily cricket powder consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutrition, Mahidol University, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No